CLINICAL TRIAL: NCT06323837
Title: A Phase II Randomized, Double-blind, Placebo-controlled Clinical Trial (RCT) to Evaluate the Ability of Mirtazapine (MZP) to Increase Methamphetamine (MA) Abstinence Among Treatment-seeking Medication for Opioid Use Disorder (MOUD) Adults
Brief Title: Mirtazapine for the Treatment of Methamphetamine Use in Opioid Use Disorder Patients Receiving Medication Assisted Treatment
Acronym: MIRROM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington State University (Other)
Responsible Party: Principal Investigator, Sterling McPherson, Vice Dean of Resarch, Washington State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20383
Record Dates: First submitted 2024-03-05; First posted 2024-03-21 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Stimulant Use Disorder
MeSH Terms: interventions — Mirtazapine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- MZP+TAU (Experimental): Mirtazapine + Treatment as Usual
  Interventions: Drug: Mirtazapine
- PLO+TAU (Placebo Comparator): Placebo + Treatment as Usual
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mirtazapine — This is a Phase 2, randomized, double-blind, placebo-controlled clinical trial (RCT) to evaluate the ability of mirtazapine (MZP) to increase methamphetamine (MA) abstinence among treatment-seeking medication for opioid use disorder (MOUD) adults.
  Arms: MZP+TAU
Drug: Placebo — Placebo to match.
  Arms: PLO+TAU

SUMMARY:
This project will evaluate the ability of Mirtazapine (MZP), a pharmacologically unique medication with a growing body of evidence to support its efficacy and safety for the treatment of methamphetamine (MA) use among medication for opioid use disorder (MOUD) patients, to significantly decrease MA use and related health-impairing behaviors. MZP has already successfully been used in the treatment of methamphetamine (detailed further below and in the Appendices).

The investigators hypothesize that those assigned to the MZP plus treatment as usual (TAU) MZP+TAU arm will demonstrate significantly increased rates of biochemically verified abstinence from MA and other substances of abuse and experience improvements in health impairing behaviors relative to the placebo (PLO)+TAU arm across the 10-week treatment and follow-up periods.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment at medication for opioid use disorder (MOUD) treatment at Oregon Recovery & Treatment Center/clinics in Spokane, WA.
* Verification of a DSM-5104 diagnosis of an methamphetamine (MA) use disorder (i.e. mild, moderate, or severe),
* Aged 18+ years,
* Ability to provide written informed consent,
* Demonstration of 78% adherence rate during the induction period and
* Provision of at least one MA positive urinalysis at baseline or during induction.
* Baseline complete blood cell count (CBC), total protein, albumin, glucose, alkaline phosphatase, creatinine, BUN, and electrolytes without clinically significant abnormalities as determined by clinician in conjunction with symptoms, physical exam, and medical history.
* No current acute illness requiring prolonged medical care.
* No serious chronic illnesses that are likely to progress clinically during trial participation.
* Vital signs are within the normal ranges (i.e., Blood pressure: 90/60 mm Hg to 120/80 mm Hg; breathing: 12-18 breaths per minute; pulse: 60-100 beats per minute; temperature: 97.8 - 99.1 degrees Fahrenheit.

Exclusion Criteria:

* Inability to demonstrate competency to provide informed consent because of cognitive or psychiatric disorders or limited English proficiency,
* Prior diagnosis of dementia,
* Medically or psychiatrically unsafe to participate as determined by Dr. Layton (Medical Director),
* Documented suicide attempt in the past 30 days and/or serious suicide intention or plan as assessed by the Structured Clinical Interview for DSM-5 (SCID-5; clinical trials version)105
* Suicide attempt in the last 2 years
* Moderate or severe liver disease (AST, ALT, and total bilirubin >= 5 times upper limit of normal),
* Impaired renal function (estimated GFR <40 ml/min),
* Current severe cocaine, amphetamine, or alcohol use disorder as defined by DSM-5 criteria which Drs Layton and McPherson deem their participation as unsafe.
* History of bipolar disorder or psychotic disorder, as determined by Structured Clinical Interview for DSM Disorders (SCID,
* Currently taking 1) any type of opioid use disorder medication other than methadone or buprenorphine/naloxone, or 2) phenytoin, carbamazepine, or another inducer of hepatic metabolism (such as rifampicin) and CYP enzyme inhibitor cimetidine.
* Taking an anti-depressant medication within the past 30 days, including mirtazapine or a monoamine oxidase inhibitor,
* Prescribed MZP in the least year, or
* History of violent criminal behavior or being on parole,.
* Currently pregnant or intending to become pregnant,.
* Final determination of eligibility will be made by Dr. Layton in consultation with the PI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-17 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Urinanalysis Verified Increased Days of MA Abstinence | Weeks 2 to Week 22
  Determine if participants randomized to the MZP+TAU arm use less MA compared to those assigned to the PLO+TAU arm. We hypothesize that those assigned to the MZP+TAU arm will demonstrate significantly increased rates of biochemically verified MA abstinence relative to those in the PLO+TAU arm across the 10-week treatment period and 3-month follow-up periods.

SECONDARY OUTCOMES:
Actigraphy Verified Improved Sleep Patterns | Week 2 to Week 22
  Determine if participants randomized to the MZP+TAU arm demonstrate improvements in sleep compared to those assigned to the PLO+TAU arm. We hypothesize that those assigned to the MZP+TAU arm will demonstrate improvements in objectively verified sleep relative to the PLO+TAU arm across the 10-week treatment and 3-month follow-up periods.

OTHER OUTCOMES:
Self Reported Quantity of Adverse Events | Week 2 to Week 22
  Determine if participants randomized to the MZP+TAU arm experience the same number of adverse events compared to those in the PLO+TAU arm. We hypothesize that those assigned to the MZP+TAU arm will demonstrate statistically equivalent numbers of adverse events relative to those in the PLO+TAU arm across the 10-week treatment and 3-month follow-up periods.
Urinanalysis Verified Increased Days of Abstinence from Other Substances | Week 2 to Week 22
  Determine if participants randomized to the MZP+TAU arm abstain from other substances of abuse (e.g. illicit opioids, cocaine) and demonstrate improvements in MA-associated health-impairing outcomes (e.g. cravings, sleep quality and HIV risk behavior) compared to those assigned to the PLO+TAU arm.

CONTACTS AND LOCATIONS:
Overall Officials: Sterling M McPherson, PhD, Principal Investigator — Washington State University
Locations (1):
- Spokane Treatment Center, Spokane, Washington, United States